CLINICAL TRIAL: NCT07378488
Title: Structured Dance/Movement Therapy for Functional Neurological Disorder: A Feasibility Study
Brief Title: Dance/Movement Therapy for Functional Neurological Disorder
Acronym: DMTforFND
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HR-25/26-51710
Record Dates: First submitted 2026-01-13; First posted 2026-01-30 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Functional Neurological Disorder
Keywords: Functional Neurological Disorder; Dance Movement Therapy; Interoception; FND; Intervention; Physical Exercise
MeSH Terms: conditions — Conversion Disorder; Motor Activity | interventions — Movement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: One research team member, leading the collection of laboratory data and inputting secondary outcome measures, will be blinded to group assignment. Participants will be reminded not to disclose information related to group allocation to this team member to prevent possible bias during the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Structured dance/movement therapy (Experimental): Participants will receive a structured dance/movement therapy programme over a period of five weeks
  Interventions: Other: Structured dance/movement
- Physical exercise/body coordination (Active Comparator): Participants will receive a physical exercise/body coordination programme over a period of five weeks
  Interventions: Other: Physical exercise/body coordination

INTERVENTIONS:
Other: Structured dance/movement — Fifteen participants will be randomly assigned using a computer-generated allocation sequence to the dance/movement intervention. This will involve a combination of light stretching, warming up using contact with a stress ball, and aerobic dance movements which follow the rhythm of a piece of music. It will be accessible to a range of abilities and will take ~30 minutes.
  This intervention has been developed with the aim of:
  * Enhancing adaptive bodily awareness, allowing the participant to feel more safe and at home in their body while promoting accurate and non-judgmental detection of bodily signals
  * Working with rhythms and coordinated movements leading to the elevation of the salience of bodily signals (heartbeat, sweating) in a structured setting - promoting adaptive noticing of signals in the body, not distracting from what one might be feeling.
  * Helping participants to engage with their body, notice and sense what they're feeling, and feel more comfortable moving their body.
  Arms: Structured dance/movement therapy
Other: Physical exercise/body coordination — Fifteen participants will be randomly assigned to this task. This will involve simple functional stretches, balances and limb coordination exercises and will use only neutral instructions. It will be accessible to a range of abilities and will take ~30 minutes.
  This task has been developed as the control condition with the following in mind:
  * Including functional movement matched for level of aerobic intensity to the dance/movement task.
  * Matching the length of the task and level of contact with the lead researcher/research team.
  * No prompts or explicit instructions to focus on bodily sensations, the self or body in the present moment, or to move in an expressive way; purely focused on mobility and physical functioning.
  Arms: Physical exercise/body coordination

SUMMARY:
Building on evidence for somatic or physical interventions in functional neurological disorder (FND), the goal of this study is to test the feasibility of a structured dance/movement task in individuals with FND, and explore the potential use of somatic or body-based therapies in this population.

The primary study outcomes will be the feasibility and acceptability of a structured dance/movement therapy (DMT) intervention for individuals diagnosed with FND. The study will also explore whether this type of intervention has potential to contribute to elevating trust in the body and general wellbeing, alongside reducing functional neurological and dissociative symptoms.

Researchers will compare structured dance/movement therapy to a physical exercise/body coordination condition.

DETAILED DESCRIPTION:
Functional neurological disorder (FND) sits in between neurology and psychiatry, including symptoms like tremors, limb weakness, functional seizures, and sensory issues. Previous research has found elevated dissociative symptoms (i.e., feelings of detachment or disconnection from the self or surroundings) and/or dissociative disorder comorbidities (i.e., dissociative identity disorder, dissociative amnesia) in FND populations relative to the general population. There is also emerging evidence for alterations in aspects of bodily awareness in FND, specifically including a lack of trust in the body and an increased tendency or likelihood to distract from bodily sensations, and atypical autonomic reactivity. These alterations may contribute to, or play a role in the experience of, FND symptoms.

Dance/movement therapy (DMT) may be a potentially beneficial intervention for disorders characterized by bodily symptoms or feelings of disconnection from the self, including FND. Generally, DMT is based on the premise that psychological and bodily experiences reciprocally influence one another and has been shown to improve health-related psychological outcomes and wellbeing in a range of populations (e.g., fibromyalgia, brain trauma). Previous research has shown promise for body-based approaches for the treatment of dissociation and trauma-related distress, encouraging individuals to attend to their bodies/bodily sensations.

Previous research demonstrates reductions in bodily disconnection post-DMT in individuals with Depersonalization-Derealization disorder, a dissociative disorder that, like FND, involves disconnections from the self and surroundings and alterations to bodily awareness (lack of trusting the body, difficulties with attention regulation). Using structured DMT for FND may help to encourage a conscious connection to the body/surroundings in the here and now, as well as a recognition of bodily states and, in turn, an adaptive regulation of them. The feasibility of dance/movement therapy has not yet been tested in FND and may provide new avenues for treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or older
* Fluency in English language
* Normal or corrected eyesight
* Primary diagnosis of FND with seizures, motor symptoms, sensory symptoms, or mixed FND symptoms
* Participants will be asked to provide proof of FND diagnosis in the form of an existing medical letter from a qualified healthcare professional (not required to be from an NHS service). This will be checked prior to engaging in the screening interview for the study.

Exclusion Criteria:

* Physical symptoms or disability that would prohibit the participant's ability to engage with the intervention and/or attend the in-person sessions (e.g., upper/lower limb paralysis, seizure frequency > 10 per day, severe tremor)
* A diagnosis of functional cognitive disorder or functional cognitive symptoms only
* Current participation in another body-based therapy or intervention for FND - participants currently engaging in some form of body- based therapy, whether self-guided or therapist-guided, will be asked to abstain from these sessions during the course of this study. If this is not feasible, the participant will be excluded from the current study.
* Current comorbid diagnosis of a major neurological (e.g., epilepsy, Parkinson's), psychiatric (e.g., schizophrenia, active psychosis, severe alcohol or substance use disorder), or cardiovascular (e.g., coronary artery disease, heart failure) disorder that may impair the participant's ability to participate in the study and confound the results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-28 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-28 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the intervention: Recruitment | Up to 16 weeks
  The number/proportion of eligible participants who consent to participate in the study by 29/05/2026
Feasibility of the intervention: Adherence | Up to 20 weeks
  The number/proportion of in-person visits and mid-point calls attended and completed. The number of days the task was completed during the at-home periods.
Feasibility of the intervention: Withdrawal | Up to 20 weeks
  The number/proportion of enrolled (consented) participants who withdraw from the study prior to completion.
Feasibility of the intervention: Adverse events | Up to 20 weeks
  The number and nature of adverse events reported during study participation.
Feasibility of the intervention: Acceptability | Up to 20 weeks
  Qualitative measures of perceived benefit of the intervention, barriers and facilitating factors, experiences of study procedures.

SECONDARY OUTCOMES:
Clinical Global Impression - Improvement Scale | Baseline, Week 2.5, Week 5, Week 9
  This is a one question measure that assesses self-reported current symptom severity relative to study intake. Patients will rate their current functional neurological disorder symptoms using this 7-point scale (1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6= much worse; 7=very much worse).
Functional Neurological Symptoms Questionnaire | Baseline, Week 2.5, Week 5, Week 9
  Measures the presence, impact, and severity of functional neurological symptoms including seizures, tremors, etc.
Multidimensional Assessment of Interoceptive Awareness - 2 | Baseline, Week 2.5, Week 5, Week 9
  A 37-item self-report questionnaire assessing various abilities relating to awareness and recognition of bodily experiences, including eight subscales: Noticing, Not-Distracting, Not- Worrying, Attention Regulation, Emotional Awareness, Self-Regulation, Body Listening, Trust. Each question is rated from 0-5, and average scores are calculated across the items for each subscale. Higher scores on all subscales indicate better outcomes.
Five Facet Mindfulness Questionnaire | Baseline, Week 2.5, Week 5, Week 9
  A 39-item scale with five facets (Observing, Describing, Acting with Awareness, Non-Judging, Non-Reactivity) measuring trait mindfulness in everyday life each facet. Each question is rated from 1-5, with higher scores indicating better outcomes.
Cognitive Behavioural Response Questionnaire - Short Form | Baseline, Week 2.5, Week 5, Week 9
  An 18-item self-report scale to capture cognitive and behavioural responses to symptoms with six subscales: Fear Avoidance, Damaging Beliefs, Embarrassment Avoidance, Symptom Focusing, All-or-Nothing Behaviour, Resting Behaviour. Each question is rated from 0-4, with higher scores across subscales indicating worse outcomes.
Multiscale Dissociation Inventory | Baseline, Week 2.5, Week 5, Week 9
  A 30-item self-report measure that assesses different types of psychological dissociative symptoms across five subscales: Disengagement, Depersonalisation, Derealisation, Memory Disturbance, Emotional Constriction, and Identity Dissociation. Each question is rated on a scale from 1-5, with total scores on each subscale (ranging from 5-25) converted into T scores once calculated. Higher scores indicate worse outcomes.
Toronto Alexithymia Scale - 20 | Baseline, Week 2.5, Week 5, Week 9
  A 20-item self-report questionnaire assessing alexithymia across a total score and three subscales: Difficulty Describing Feelings, Difficulty Identifying Feelings, Externally Oriented Thinking. Total scores range from 20-200, with higher scores indicating worse outcomes.
Work & Social Adjustment Scale | Baseline, Week 2.5, Week 5, Week 9
  A five-item self-report measure assessing impairments in social and occupational functioning. Total scores range from 0-40, with higher scores indicating worse outcomes.
Short-Form Health Survey | Baseline, Week 2.5, Week 5, Week 9
  A 36-item measure of health-related quality-of-life over the past four weeks across eight subscales: Physical Functioning, Role Limitations Due to Physical Health, Role Limitations Due to Emotional Problems, Energy and Fatigue, Emotional Wellbeing, Social Functioning, Pain, and General Health. Individual items are rated from 1-6 and, after participant ratings, each item is recoded on a 0-100 scale, with higher scores indicating better outcomes.
Body Perception Questionnaire - ANS | Baseline, Week 2.5, Week 5, Week 9
  A 20-item scale measuring autonomic nervous system symptoms in everyday life. Total scores range from 20-100, with higher scores indicating worse outcomes.
Body Perception Questionnaire - VSF | Baseline, Week 2.5, Week 5, Week 9
  A 12-item scale measuring awareness of particular sensations within the body. Total scores range from 12-60, with higher scores indicating greater sensitivity to internal bodily sensations.
Cardiac interoceptive accuracy | Day 1 baseline, Day 1 post single intervention session, Week 5
  Measured using a heartbeat tracking task (HTT) in the laboratory. Participants are asked to pay attention to and count the number of heartbeats they feel over different periods of time to determine how accurate they are with regards to this, over four trials.
Cardiac interoceptive confidence | Day 1 baseline, Day 1 post single intervention session, Week 5
  Measured using a heartbeat tracking task (HTT) in the laboratory. Participants are asked to judge their level of confidence in how accurate the are in detecting their heartbeats over four trials within the task.
Time estimation accuracy | Day 1 baseline, Day 1 post single intervention session, Week 5
  A control task to the heartbeat tracking task (HTT) where participants are asked to count seconds over differing periods of time to measure their accuracy with regards to time perception, over four trials.
Time estimation confidence | Day 1 baseline, Day 1 post single intervention session, Week 5
  A control task to the heartbeat tracking task where participants are asked to count seconds over differing periods of time to, indicating their confidence in this ability over four trials.
Physiological and psychological states | Day 1 baseline, Day 1 post single intervention session, Week 5
  Measured in the laboratory. Self-report questions of current state pain, bodily/autonomic arousal, fatigue, functional neurological symptoms, and dissociation.
Autonomic arousal | Day 1 baseline, Day 1 post single intervention session, Week 5
  Participants will be asked to wear sensors to measure their heartrate and electrical conductivity of the skin (measures of physiological/autonomic arousal). Heartrate will be measured with electrocardiography: two sensors will be attached under the collarbones and one on the left ankle. Electrical conductivity of the skin/electrodermal activity will be measured with two sensors on the index and middle fingers of the non- dominant hand. The electrocardiography sensors will also be worn during completion of the heartbeat tracking and time estimation tasks.
At-home Diary Sheet: ease of task performance | Day 3, Day 6, Day 9, Day 12, Day 15, Day 18, Day 21, Day 24, Day 27, Day 30
  Completed on days when participants perform the intervention or control task at home. Post task, participants are asked to indicate on a 1-7 Likert scale (1: very easy, 7: very difficult) how easy it was to perform the task.
At-home Diary Sheet: feeling during task performance | Day 3, Day 6, Day 9, Day 12, Day 15, Day 18, Day 21, Day 24, Day 27, Day 30
  Completed on days when participants perform the intervention or control task at home. Post task, participants are asked to indicate on a 1-7 Likert scale (1: very bad, 7: very good) how they felt while performing the task.
At-home Diary Sheet: physical states | Day 3, Day 6, Day 9, Day 12, Day 15, Day 18, Day 21, Day 24, Day 27, Day 30
  Completed on days when participants perform the intervention or control task at home. Likert scale from 1-7 (1: not at all, 7: extremely) measuring current state: pain, bodily arousal, fatigue, functional neurological symptoms (e.g., tremors, weakness, seizures, tingling/numbness).
At-home Diary Sheet: state dissociation | Day 3, Day 6, Day 9, Day 12, Day 15, Day 18, Day 21, Day 24, Day 27, Day 30
  Completed on days when participants perform the intervention or control task at home. Ten questions of state dissociation (e.g., feeling detached from oneself and surroundings) from the Clinician Administered Dissociative States Scale, measured on a scale from 0 (not at all) to 4 (extremely) and total scores ranging from 0-40.
At-home Diary Sheet: autonomic arousal | Day 3, Day 6, Day 9, Day 12, Day 15, Day 18, Day 21, Day 24, Day 27, Day 30
  Completed on days when participants perform the intervention or control task at home. Post task, two questions regarding the ability to currently feel one's heartbeat (yes/no) and if one is currently sweating (yes/no).
At-home Diary Sheet: open comments | Day 3, Day 6, Day 9, Day 12, Day 15, Day 18, Day 21, Day 24, Day 27, Day 30
  Completed on days when participants perform the intervention or control task at home. Open comments box for participants to add any thoughts or feelings about the session.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Psychiatry, Psychology and Neuroscience, King's College London, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
The datasets of the study will be available from the corresponding author on reasonable request after the findings have been published in relevant peer-reviewed journals.

REFERENCES:
- [Background] Kennedy-Barnes E, Millman LSM, Basamh Y, Duarte A, Pacelli J, Hodsoll J, Pick S. Somatic yoga therapy for functional neurological disorder: A feasibility randomised controlled trial. https://doi.org/10.31234/osf.io/r3cgf_v1
- [Background] Pick S, Rojas-Aguiluz M, Butler M, Mulrenan H, Nicholson TR, Goldstein LH. Dissociation and interoception in functional neurological disorder. Cogn Neuropsychiatry. 2020 Jul;25(4):294-311. doi: 10.1080/13546805.2020.1791061. Epub 2020 Jul 8. PMID 32635804
- [Background] Pick S, Goldstein LH, Perez DL, Nicholson TR. Emotional processing in functional neurological disorder: a review, biopsychosocial model and research agenda. J Neurol Neurosurg Psychiatry. 2019 Jun;90(6):704-711. doi: 10.1136/jnnp-2018-319201. Epub 2018 Nov 19. PMID 30455406
- [Background] Millman LSM, Hunter ECM, Terhune DB, Orgs G. Online structured dance/movement therapy reduces bodily detachment in depersonalization-derealization disorder. Complement Ther Clin Pract. 2023 May;51:101749. doi: 10.1016/j.ctcp.2023.101749. Epub 2023 Mar 30. PMID 37018935
- [Background] Millman LSM, Short E, Stanton B, Winston JS, Nicholson TR, Mehta MA, Reinders AATS, Edwards MJ, Goldstein LH, David AS, Hotopf M, Chalder T, Pick S. Interoception in functional motor symptoms and functional seizures: Preliminary evidence of intact accuracy alongside reduced insight and altered sensibility. Behav Res Ther. 2023 Sep;168:104379. doi: 10.1016/j.brat.2023.104379. Epub 2023 Jul 25. PMID 37516011